CLINICAL TRIAL: NCT06295653
Title: Subepithelial Connective Tissue Graft Versus Amniotic Chorion Membrane for Peri-implant Mucosal Thickness Enhancement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Hamdy Helal, Lecturer of Oral Medicine, Periodontology, Oral Diagnosis & Radiology, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 7-23
Record Dates: First submitted 2023-09-21; First posted 2024-03-06 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Dental Implant
Keywords: dental implant; Subepithelial Connective Tissue Graft; Amniotic Chorion Membrane; for Peri-implant Mucosa

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous Subepithelial Connective Tissue Graft plus dental implants (Active Comparator): implant placement and augment Subepithelial Connective Tissue Graft and suture implant site
  Interventions: Procedure: implant placement and soft tissue augmentation with Autogenous Subepithelial Connective Tissue Graft or Amniotic Chorion Membrane
- Amniotic Chorion Membrane plus dental implant (Active Comparator): implant placement and augment Amniotic Chorion Membrane and suture implant site
  Interventions: Procedure: implant placement and soft tissue augmentation with Autogenous Subepithelial Connective Tissue Graft or Amniotic Chorion Membrane

INTERVENTIONS:
Procedure: implant placement and soft tissue augmentation with Autogenous Subepithelial Connective Tissue Graft or Amniotic Chorion Membrane — assess the efficacy of the peri-implant mucosal thickness enhancement following either subepithelial connective tissue grafts or Amniotic Chorion Membrane placed simultaneously with dental implant placement.
  Other Names: measure mucosal thickness with probe; connective tissue grafting from palate

SUMMARY:
The objective of this study will be to assess the efficacy of the peri-implant mucosal thickness enhancement following either subepithelial connective tissue grafts or Amnion Chorion Membrane placed simultaneously with dental implant placement.

ELIGIBILITY:
Inclusion Criteria:

* Patients with good systemic health with no contraindication for periodontal surgery.
* No history of any medications in the previous 6 months that may interfere with periodontal tissue health or healing.
* Ability to maintain good oral hygiene as evidenced in recall visits.
* Aged 30 to 55 years.
* Stable periodontal condition and missing one single tooth (maxillary anterior teeth and premolars) with adjacent teeth present and thin mucosal phenotype (< 2mm bucco- lingual thickness).

Exclusion Criteria:

* Medically compromised patients and systemic conditions precluding periodontal surgery.
* Smokers.
* Severe hematologic disorders (e.g., hemophilia or leukemia), uncontrolled infectious or metabolic diseases that could compromise normal healing, liver, or kidney dysfunction/failure.
* Patients subjected to irradiation in the head and neck area.
* Patients treated or under treatment with intravenous amino bisphosphonates.
* Patient affected by active periodontitis or has poor oral hygiene and motivation.
* Uncontrolled diabetes mellitus.
* Pregnant women or planning become pregnant, and nursing mothers.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2024-04-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
measure changes in periimplant mucosal thickness | six months
  The primary outcome of interest will be to measure changes (in mm) in horizontal periimplant mucosal thicknesson the buccal aspect of the edentulous alveolar ridge from baseline (BL) (implant placement and grafting) to (3 and 6 month) of post-surgical healing.

SECONDARY OUTCOMES:
mid-buccal keratinized mucosal width | six month
  measure change (in mm) in mid-buccal keratinized mucosal width in an apico-coronal direction

CONTACTS AND LOCATIONS:
Locations (1):
- Faculity of Dentistry Tanta University, Tanta, Elgarbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
share the results to determine the difference between the materials used in the research and the possibility of using the best ones
Supporting Information: SAP
Time Frame: at the end of the research When the data are available

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-03-03): https://cdn.clinicaltrials.gov/large-docs/53/NCT06295653/Prot_SAP_000.pdf